CLINICAL TRIAL: NCT06651138
Title: A Single-Center Prospective Study Evaluating Efficacy of Radiation Exposure Reduction Protocol for Minimally Invasive Lumbar Decompression (mild) Techniques Including Single Incision Access
Brief Title: Radiation Exposure Reduction Protocol for Minimally Invasive Lumbar Decompression (mild) Techniques
Status: Withdrawn | Type: Observational
Why Stopped: Study did not move forward at our institution
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Dawood Sayed, MD, Study Principal Investigator, University of Kansas Medical Center
Other Study IDs: STUDY00145205
Record Dates: First submitted 2020-12-22; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Spinal Stenosis; Radiation Exposure
Keywords: fluoroscopy; radiation exposure reduction; Minimally Invasive Lumbar Decompression
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs and hypertrophic tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pulsed Fluoroscopy: Patients in the study group will receive pulsed (8 frames/second) fluoroscopy for the entirety of the procedure
  Interventions: Radiation: Fluoroscopy
- Continuous Fluoroscopy: Non-study arm patients will receive continuous fluoroscopy for the entire procedure
  Interventions: Radiation: Fluoroscopy

INTERVENTIONS:
Radiation: Fluoroscopy — Pulsed or Continuous fluoroscopy during MILD procedure

SUMMARY:
To evaluate the efficacy of radiation reduction techniques to minimize clinician and patient exposure during minimally invasive lumbar decompression (MILD) procedure. Additionally, to evaluate the clinical benefits of single incision access for bilateral mild procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years old
* Patient has meets eligibility criteria for (mild)
* Patient has signed study-specific informed consent form
* Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements
* Patient has medical insurance that covers this standard of care procedure and all other anticipated and unanticipated procedure related care.

Exclusion Criteria:

* Patient does not meet criteria for mild
* Patient is unable to receive radiation exposure.
* Current local or systemic infection that raises the risk of surgery
* Patient currently receiving or seeking worker's compensation, disability remuneration, and/or involved in injury litigation.
* Currently pregnant
* Known or suspected drug or alcohol abuse
* Diagnosed psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation
* Patient is participating in an investigational study or has been involved in an investigational study within 3 months prior to evaluation for participation
* Implanted intrathecal pain pump or spinal cord stimulator system in place
* Patient who has received other means pain management with minimally invasive implantable devices (spacer, sacroiliac joint (SIJ) fusion, etc).
* Patient with physical inability to ambulate independently, otherwise.
* Patient underlying neurologic pathology preventing safe independent ambulation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Individuals 65 years or older experiencing lumbar spinal stenosis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Pulsed fluoroscopy can reduce radiation exposure to clinicians and patients compared to continuous fluoroscopy | During surgery
  Compare patient outcome in the study group receiving pulsed (8 frames/second) fluoroscopy for the entirety of the procedure to non-study arm patients who will receive continuous fluoroscopy for the entire procedure.
Genetic factors can explain individual differences in pain severity and the response to MILD (with and without pulsed fluoroscopy) | Up to 6 months post-surgery
  We will store, run and analyze buccal cell samples for pain-related genetic variations (polymorphisms). Buccal cell samples will be collected at baseline/time of recruitment for this study.

SECONDARY OUTCOMES:
Average rate of complications | During surgery
  Average rate of complications is comparable for Pulsed fluoroscopy from mild procedure compared to continuous fluoroscopy
Duration of surgery | During surgery
  Compare difference in duration of the mild procedure utilizing Pulsed fluoroscopy compared to continuous fluoroscopy.
Patient BMI | During surgery
  Compare use of pulsed fluoroscopy depending on patient BMI
Difference in average Visual Analogue Scale (VAS) | Up to 6 months post-treatment
  Compare difference in average VAS between Pulsed fluoroscopy and continuous fluoroscopy post mild procedure
Single Nucleotide Polymorphisms (SNPs) within pain-relevant genes will be predictive of pre-surgical pain severity prior to MILD | Up to 6 months post-treatment
  Compare genetic expression profile to pain severity self report pre surgery
Single Nucleotide Polymorphisms (SNPs) within pain and/or analgesia relevant genes will be predictive of pain relief following MILD (with continuous or pulsed fluoroscopy). | Up to 6 months post-treatment
  Compare genetic expression profile to pain severity self report post surgery
Establish patient "profile of risk" | Up to 6 months post-treatment
  The pattern of gene expression (i.e. the transcriptome) within lumbar hypertrophic tissue can be used to establish a patient "profile of risk" for pre-surgical pain severity, pain relief response to MILD, and recurrence of hypertrophic tissue following the MILD procedure (with continuous or pulsed fluoroscopy).

CONTACTS AND LOCATIONS:
Overall Officials: Dawood Sayed, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States